CLINICAL TRIAL: NCT02589626
Title: A 52-week Randomised, Double-blind, Parallel Group, Safety and Efficacy Study of Empagliflozin Once Daily as add-on Therapy to Glucagon-like Peptide-1 Receptor Agonist in Japanese Type 2 Diabetes Mellitus Patients With Insufficient Glycaemic Control
Brief Title: Long-term Safety and Efficacy of Empagliflozin as Add on to GLP-1 RA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.106
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (2):
- empagliflozin 10 mg (Experimental): empagliflozin 10 mg tablet and placebo matching empagliflozin 25 mg tablet
  Interventions: Drug: empagliflozin 10mg; Drug: Placebo
- empagliflozin 25 mg (Experimental): empagliflozin 25 mg tablet and placebo matching empagliflozin 10 mg tablet
  Interventions: Drug: empagliflozin 25 mg; Drug: Placebo

INTERVENTIONS:
Drug: empagliflozin 10mg
  Arms: empagliflozin 10 mg
Drug: empagliflozin 25 mg
  Arms: empagliflozin 25 mg
Drug: Placebo — For blinding purposes

SUMMARY:
This is a multi-center, randomised, double-blind, parallel-group, safety and efficacy study of empagliflozin as add-on to GLP-1 RA in Japanese patients with Type 2 Diabetes Mellitus with insufficient glycaemic control

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of type 2 diabetes mellitus
* Male and female patients on diet and exercise regimen who are pre-treated with Liraglutide at 0.9 mg/day alone for at least 10 weeks prior to screening must be >=7.0% and <=10.0% at screening
* Male and female patients on diet and exercise regimen who are pre-treated with Liraglutide at 0.9 mg/day and one of oral antidiabetic drug (OAD) for at least 10 weeks prior to Visit 1 must be >=7.0% and <=9.0% at screening and >=7.0% and <=10.0% at placebo run-in
* Male and female patients on diet and exercise regimen who are pre-treated with OAD alone for at least 10 weeks prior to Visit 1 must be >=7.0% and <=10.0% at both screening and placebo run-in
* Age at informed consent must be >=20 years
* BMI at screening must be <=40 kg/m2
* Further inclusion criteria apply

Exclusion criteria:

* Uncontrolled hyperglycaemia with a glucose values >270 mg/dL (>15.0 mmol/L) after an overnight fast during switch/washout/placebo run-in period and confirmed by a second measurement
* Patients who are drug-naïve at screening visit or treat with any of insulin, thiazolidine dione, sodium-glucose co-transporter 2 (SGLT-2) inhibitor within 10 weeks prior to informed consent.
* Acute coronary syndrome, stroke or transient ischemic attack within 12 weeks prior to informed consent
* Indication of liver disease, defined by serum levels of either alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase above 3 x upper limit of normal as determined during screening and/or switch/washout/placebo run-in period
* Impaired renal function, defined as estimated glomerular filtration rate (eGFR) <45 mL/min/1.73m2 (Japanese equation) as determined during screening and/or switch/washout/placebo run-in period
* Further exclusion criteria apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (16):
- Japan (16):
  - Kunisaki Makoto Clinic, Fukuoka, Fukuoka
  - Seino I.M. Clinic, Fukushima, I.M., Fukushima, Koriyama
  - Nippon Kokan Fukuyama Hospital, Hiroshima, Fukuyama
  - Nakakinen Clinic, Ibaraki, Naka
  - Kubota Clinic, Kanagawa, Kawasaki
  - Medical Corporation Yuga Higashirinkan Kaneshiro Diabetes Clinic, Kanagawa, Yamato-shi
  - Yokohama Minoru Clinic, Kanagawa, Yokohama
  - Yokkaichi Diabetes Clinic, Mie, Yokkaichi
  - Shiraiwa Medical Clinic, Osaka, Kashiwara-shi
  - AMC Nishi-umeda Clinic, Osaka, Osaka-shi
  - OCROM Clinic, Osaka, Suita
  - Fukuwa Clinic, Tokyo, Chuo-ku
  - Tokyo-Eki Center-building Clinic, Tokyo, Chuo-ku
  - Minamino Heart Clinic, Tokyo, Hachioji
  - ToCROM Clinic, Tokyo, Shinjuku-ku
  - Shinjuku Research Park Clinic, Tokyo, Shinjuku-ku

REFERENCES:
- [Derived] Terauchi Y, Utsunomiya K, Yasui A, Seki T, Cheng G, Shiki K, Lee J. Safety and Efficacy of Empagliflozin as Add-On Therapy to GLP-1 Receptor Agonist (Liraglutide) in Japanese Patients with Type 2 Diabetes Mellitus: A Randomised, Double-Blind, Parallel-Group Phase 4 Study. Diabetes Ther. 2019 Jun;10(3):951-963. doi: 10.1007/s13300-019-0604-8. Epub 2019 Mar 25. PMID 30912033

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were entered in the trial and randomised in a 1:1 ratio to receive treatment.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist site which would then ensure that they (the subjects) met all strictly implemented inclusion/exclusion criteria. Subjects were not randomised to trial treatment if any one of the specific entry criteria was violated.
Groups:
- Empagliflozin 10 mg: Patients were orally administered film-coated tablet of Empagliflozin 10 milligram (mg) once daily in the morning for 52 weeks
- Empagliflozin 25 mg: Patients were orally administered film-coated tablet of Empagliflozin 25 mg once daily in the morning for 52 weeks
Period: Overall Study
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg
Started | 32 (Entered are treated patients) | 33 (Entered are treated patients)
Completed | 29 | 31
Not Completed | 3 | 2
Not completed — Other than the reason specified | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set:
  The full analysis set (FAS) consisted of all patients in the treated set (TS) who were treated with at least 1 dose of the randomised study drug and had a baseline HbA1c assessment. The assignment of patients to treatment groups was based on the randomised study drug at time of randomisation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Full analysis set The full analysis set (FAS) consisted of all patients in the TS who were treated with at least 1 dose of the randomised study drug and had a baseline HbA1c assessment. The assignment of patients to treatment groups was based on the randomised study drug at time of randomisation.
  years | 55.6 (9.8) | 58.9 (9.3) | 57.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Female | 6 | 11 | 17
    Male | 26 | 22 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: FAS
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 32 | 33 | 65
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Baseline glycosylated haemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: % of HbA1c] — Population: FAS
  % of HbA1c | 8.83 (0.80) | 8.68 (0.87) | 8.76 (0.83)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Drug-related Adverse Events (AEs) During 52 Weeks of Treatment
Description: Percentage of patients with drug-related Adverse events (AEs) during 52 weeks of treatment are presented
Time Frame: 52 weeks
Population: The treated set (TS) consisted of all patients who were randomised and treated with at least 1 dose of the study drug. The assignment of patients to treatment group was based on the first study drug intake in the double-blind treatment period.
Measure: Number; unit: Percentage of participants
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 32 | 33
Percentage of participants | 9.4 | 21.2

2. Secondary Outcome: Change From Baseline in HbA1c After 52 Weeks of Treatment
Description: Change from baseline in HbA1c after 52 weeks of treatment is presented. Means presented are the adjusted means.
Time Frame: baseline and 52 weeks
Population: Full Analysis Set (Observed cases (OC))
Measure: Mean (Standard Deviation); unit: % of HbA1c
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 32 | 33
% of HbA1c | -0.55 (0.15) | -0.77 (0.14)

ADVERSE EVENTS:
Time Frame: All AEs which occurred through the treatment phase and throughout the residual effect period (REP); up to 53 weeks
Groups:
- Empagliflozin 25mg: Patients were orally administered film-coated tablet of Empagliflozin 10 mg once in the morning for 52 weeks
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25mg
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 2/32 | 1/33
Other Adverse Events (participants affected / at risk) | 10/32 | 15/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 10 mg (N=32) | Empagliflozin 25mg (N=33)
Loss of consciousness (Nervous system disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 10 mg (N=32) | Empagliflozin 25mg (N=33)
Viral upper respiratory tract infection (Infections and infestations) | 10 | 11
Influenza (Infections and infestations) | 0 | 3
Periodontitis (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 2
Vulvovaginal candidiasis (Infections and infestations) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property right

DOCUMENTS (2):
  • Study Protocol (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT02589626/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT02589626/SAP_001.pdf